CLINICAL TRIAL: NCT05231148
Title: Hardware Preservation in Management of Infected Non United or Delayed United Fractures of Long or Short Bones by Debridement and Local Calcium Sulfate Loaded by Antibiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelraheem Mohamed Sonbol, Resident of orthopedic surgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-01-01
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Infected Non Union and Delayed Union in Fractures of Both Long and Short Bones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infected non united fractures (Other): patient of any age and any sex with infected non united fractures of long or short bones
  Interventions: Procedure: local debridement and local calcium sulfate loaded by antibiotics

INTERVENTIONS:
Procedure: local debridement and local calcium sulfate loaded by antibiotics — debridement of infected non united fractures and placement of local calcium sulfate loaded by antibiotic then follow up at regular intervals

SUMMARY:
* Diagnosis of infection based on elevated serum markers of infection (ESR, CRP), discharging sinus, preoperative radiographs suggestive of bone infection and radiological findings . [6]
* infected nonunion mean the bone has previous fracture , the bone not healed may be one of the reasons it didn't heal because there is sub-acute infection , there is low grade colonization into the bone or around the wound preventing the bone from healing , it different from infected fracture which occur fairly acutely. [6, 7]
* Infected nonunion treated with systemic antibiotics alone, without using local antibiotic delivery systems associated with higher recurrence and reoperation rates. [7]
* This led to the development and use of medical-grade calcium sulfate (CS), CS facilitates osseous healing in an osteoconductive fashion by filling the bone void and preventing fibrous tissue

ELIGIBILITY:
Inclusion Criteria:

* Patient at any age and of any sex with infected non united fracture of long or short bones

Exclusion Criteria:

* Presence of previous vascular injury or pathological fracture
* Refusal to participate
* Inability to provide informed consent
* Allergy or sensitivity to vancomycin or tobramycin
* Patient with impaired renal function
* Patient with hypercalcemia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Non union scoring system | one year
  Non-Union Scoring System (NUSS) aims to classify non-unions according to their severity and relate them to four treatment categories.
Karlström-Olerud physical function scale | one year
  Karlström-Olerud physical function scale is a scale to assess physical functional outcome postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Calori GM, Mazza EL, Mazzola S, Colombo A, Giardina F, Romano F, Colombo M. Non-unions. Clin Cases Miner Bone Metab. 2017 May-Aug;14(2):186-188. doi: 10.11138/ccmbm/2017.14.1.186. Epub 2017 Oct 25. PMID 29263731
- [Background] Drosos GI, Ververidis A, Babourda EC, Kakagia D, Verettas DA. Calcium sulfate cement in contained traumatic metaphyseal bone defects. Surg Technol Int. 2012 Dec;22:313-9. PMID 23109071
- [Background] Laycock PA, Cooper JJ, Howlin RP, Delury C, Aiken S, Stoodley P. In Vitro Efficacy of Antibiotics Released from Calcium Sulfate Bone Void Filler Beads. Materials (Basel). 2018 Nov 13;11(11):2265. doi: 10.3390/ma11112265. PMID 30428581